CLINICAL TRIAL: NCT00280813
Title: Treatment of Alcohol Use Disorders in Schizophrenia
Brief Title: Alcohol Use Disorders in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Melanie Bennett, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21942
Record Dates: First submitted 2006-01-19; First posted 2006-01-23 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Schizophrenia; Mood Disorders; Alcohol Abuse; Alcohol Dependence
Keywords: treatment; dual diagnosis
MeSH Terms: conditions — Schizophrenia; Mood Disorders; Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Supportive Treatment in Alcohol Recovery (STAR) (Active Comparator)
  Interventions: Behavioral: Supportive Treatment in Addiction Recovery (STAR)

INTERVENTIONS:
Behavioral: Supportive Treatment in Addiction Recovery (STAR)

SUMMARY:
The purpose of the study is to evaluate a new treatment to help patients who have problems because of their use of alcohol. The treatment is called Behavioral Treatment for Alcohol Abuse in Schizophrenia (BTAAS).We are interested in determining whether BTAAS is more effective in reducing use than a supportive control treatment.

DETAILED DESCRIPTION:
Alcohol abuse and dependence in people with schizophrenia is a serious public health problem that is associated with poor treatment compliance, increased rates of relapse, increased levels of violence, and poor overall health and life functioning. Treating alcohol use disorders in people with schizophrenia is especially problematic, as schizophrenia is marked by symptoms and neurocognitive and psychosocial deficits that make it difficult for patients to engage in the higher level cognitive processes or the sustained, self-directed behaviors generally required to reduce drinking. To date there are no interventions for alcohol use disorders with solid empirical support that have been designed for or adapted to meet the needs of this multiply-handicapped population. In this study we will develop and pilot test a multifaceted behavioral intervention for treating schizophrenia patients with alcohol use disorders that will incorporate strategies that have been found to be effective in reducing drinking, but tailor them to meet the needs of this population. The intervention will contain several components, including: (1) pre-treatment motivational interviewing to increase engagement and motivation; (2) short-term goal setting at each session; (3) social skills and alcohol refusal skills training; (4) education and coping skills training for managing depression, stress and other forms of negative affect; (5) relapse prevention training; (6) case management aimed at networking with social supports in the participant's environment and linking patients with activities and social networks in the community in order to create a reinforcing, non-drinking environment.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia or schizoaffective disorder OR other severe disorder including bipolar disorder, major depression, or severe anxiety disorder (by definition, the patient has worked 25% or less of the past year; and/or the patient received payment for mental disability)
* Current (last month) Alcohol Abuse or Dependence or Alcohol Abuse or Dependence criteria met within the last 3 months as determined by the Structured Clinical Interview for DSM-IV.
* Ability to provide informed consent
* Stable housing

Exclusion Criteria:

* Current neurological disorder or cognitive impairment due to head injury or loss of consciousness that would impact ability to effectively participate in the intervention
* Mental retardation as indicated by chart review
* inability to effectively participate in the baseline assessments due to intoxication or psychiatric symptoms on two successive appointments
* patient is homeless.
* Inability to attend scheduled treatment sessions on a regular basis for any reason, or to appropriately participate in research activities due to behavioral or psychiatric problems.

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2004-03; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Symptom ratings, addiction severity, quality of life, social functioning & motivation to change: baseline and post-treatment. | 1 year

SECONDARY OUTCOMES:
Saliva test & Urinalysis: baseline, post-treatment and at each treatment session. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Bennett, Ph.D., Principal Investigator — University of Maryland, Baltimore
Locations (4):
- United States (4):
  - Healthcare for the Homeless, Baltimore, Maryland
  - University of Maryland, Baltimore, Baltimore, Maryland
  - VA Maryland Healthcare System, Baltimore, Maryland
  - Mosaic Community Services Inc., Catonsville, Maryland

REFERENCES:
- [Background] Bellack AS, DiClemente CC. Treating substance abuse among patients with schizophrenia. Psychiatr Serv. 1999 Jan;50(1):75-80. doi: 10.1176/ps.50.1.75. PMID 9890583
- [Background] Bellack AS, Gearon JS. Substance abuse treatment for people with schizophrenia. Addict Behav. 1998 Nov-Dec;23(6):749-66. doi: 10.1016/s0306-4603(98)00066-5. PMID 9801714
- [Background] Bennett ME. Interrelationship of substance abuse and mental health problems. In Miller WR & Weisner C (Eds.), Changing substance abuse through health and social systems. New York: Kluwer/Plenum, 2003.
- [Background] Bennett ME, Barnett, B.Adult psychopathology and diagnosis: Dual-diagnosis. In M. Hersen & SM Turner (Eds), Adult psychopathology and diagnosis, fourth edition. NY: Kluwer/Plenum, 2003.
- [Background] Bennett ME, Bellack AS, Gearon JS. Treating substance abuse in schizophrenia. An initial report. J Subst Abuse Treat. 2001 Mar;20(2):163-75. doi: 10.1016/s0740-5472(00)00167-7. PMID 11306219
- [Background] Miller WR, Andrews, NA, Wilbourne P, Bennett ME (1998). A wealth of alternatives: Effective treatments for alcohol problems. In Miller WR and Healther N. (Eds.). Treating addicting behaviors, second edition. NY: Plenum Press, 1998.